CLINICAL TRIAL: NCT00679432
Title: Efficacy and Safety of New Oral Budesonide-MMX™ (CB-01-02) 6 mg and 9 mg Extended Release Tablet Formulations in Patients With Mild or Moderate, Active Ulcerative Colitis. A Multicenter, Randomized, Double-blind, Double Dummy Comparative Study Versus Placebo, With an Additional Reference Arm Evaluating Asacol® 2400 mg.
Brief Title: (CB-01-02/01) Randomized Placebo Controlled Trial of Budesonide-multi-matrix System (MMX™) 6 mg and 9 mg in Patients With Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CB-01-02/01
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Results first posted 2014-08-01 (Estimated); Last update posted 2019-12-10 (Actual); Status verified 2019-11

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Blood Specimen Collection; Endoscopy; Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1: budesonide-MMX® 6 mg (Experimental): One budesonide-MMX® 6 mg plus two placebo Asacol® overencapsulated tablets daily in the morning after breakfast and two placebo Asacol® overencapsulated tablets daily after the mid-day meal and the evening meal for eight weeks.
  Interventions: Procedure: Blood sampling, endoscopy; Drug: budesonide-MMX® 6 mg
- 2: budesonide-MMX® 9 mg (Experimental): One budesonide-MMX® 9 mg plus two placebo Asacol® overencapsulated tablets daily in the morning after breakfast and two placebo Asacol® overencapsulated tablets daily after the mid-day meal and the evening meal for eight weeks.
  Interventions: Procedure: Blood sampling, endoscopy; Drug: budesonide-MMX® 9 mg
- 3: Placebo (Placebo Comparator): Two placebo Asacol® overencapsulated tablets plus one placebo Budesonide MMX® tablet daily in the morning after breakfast and two placebo Asacol® overencapsulated tablets daily after the mid-day meal and the evening meal for eight weeks.
  Interventions: Procedure: Blood sampling, endoscopy; Drug: Placebo
- 4: Asacol® 400 mg (Active Comparator): Two Asacol® 400 mg overencapsulated tablets plus one placebo budesonide MMX® tablet daily in the morning after breakfast and two Asacol® 400 mg overencapsulated tablets daily after the mid-day meal and the evening meal for eight weeks.
  Interventions: Procedure: Blood sampling, endoscopy; Drug: Asacol® 400 mg

INTERVENTIONS:
Procedure: Blood sampling, endoscopy — Blood sampling for hematology and biochemistry and endoscopy with biopsy for histological and endoscopic assessment scores
Drug: budesonide-MMX® 6 mg — 6 mg/day, 6 mg tablets
  Arms: 1: budesonide-MMX® 6 mg
Drug: budesonide-MMX® 9 mg — 9 mg/day, 9 mg tablets
  Arms: 2: budesonide-MMX® 9 mg
Drug: Placebo — Placebo
  Arms: 3: Placebo
Drug: Asacol® 400 mg — 2400 mg/day, 400 mg tablets
  Arms: 4: Asacol® 400 mg

SUMMARY:
The purpose of this study is to compare Budesonide MMX™ 6 mg and Budesonide MMX™ 9 mg tablets to placebo and to Asacol 6x 400 mg tablets over an 8-week treatment period to determine if Budesonide MMX™ is effective in the treatment of ulcerative colitis.

DETAILED DESCRIPTION:
Each patient will receive one of the following regimens in the morning after breakfast:

1. one budesonide-MMX™ 6 mg tablet plus two placebo Asacol® over encapsulated tablets, or
2. one budesonide-MMX™ 9 mg tablet plus two placebo Asacol® over encapsulated tablets, or
3. two placebo Asacol® over encapsulated tablets plus one placebo budesonide tablet, or
4. two Asacol® 400 mg over encapsulated tablets plus one placebo budesonide tablet, daily for 8 weeks.

Each patient will also receive on each day after the midday meal and after the evening meal either:

* two Asacol® 400 mg over-encapsulated tablets (Group 4), or
* the equivalent placebo Asacol® over-encapsulated tablets, (Groups 1, 2 and 3)

Hence, each patient is to take seven tablets per day of active or placebo study medication as per the randomization schedule. Placebo tablets of budesonide-MMX™ and placebo over-encapsulated tablets of Asacol® will be used to maintain the study blind using a double-dummy technique.

During the study, five visits to the clinical center are scheduled: one at Screening and three in the double-blind treatment period (Day 1, Day 14, Day 28 and Day 56). A safety follow up visit will take place about 2 weeks after the final study visit. If a patient is withdrawn from the study before Day 56, they will be asked to attend the study center as soon as possible thereafter so that the Final visit assessments can be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling the following criteria at the screening visit are eligible for participation in the study:

  * Male and female patients, 18-75 years old, suffering from ulcerative colitis for at least 6 months.
  * Diagnosis of ulcerative colitis in active phase, of mild or moderate entity with Ulcerative Colitis Disease Activity Index (UCDAI) ≥ 4 and ≤ 10 according to Sutherland.
  * All females of child-bearing potential must have a negative serum pregnancy test immediately prior to enrollment. In addition, all females of child-bearing potential must agree to be completely abstinent or be using an accepted form of contraception throughout the entire study period. Accepted forms of contraception are defined as those with a failure rate <1% when properly applied and include: combination oral pill, some intra-uterine devices, and a sterilised partner in a stable relationship. Female subjects must also not be actively breast-feeding through the entire study period.
  * Ability to comprehend the full nature and purpose of the study, including possible risks and side effects.
  * Ability to co-operate with the investigator and to comply with the requirements of the entire study.
  * Must be able to understand and voluntarily sign written informed consent prior to inclusion in the study.

Exclusion Criteria:

* Patients who meet any of the following criteria at screening visit are to be excluded from study participation:

  * Patients with limited distal proctitis (from anal verge up to 15 cm above the pectineal line).
  * Patients with severe ulcerative colitis (UCDAI >10).
  * Patients with infectious colitis.
  * Evidence or history of toxic megacolon.
  * Severe anemia, leucopenia or granulocytopenia.
  * Use of oral or rectal steroids in the last 4 weeks.
  * Use of immuno-suppressive agents in the last 8 weeks before the study.
  * Use of anti tumor necrosis factor alpha (anti-TNFα) agents in the last 3 months.
  * Concomitant use of any rectal preparation.
  * Concomitant use of antibiotics.
  * Concurrent use of cytochrome P450 3A4 (CYP3A4) inducers or CYP3A4 inhibitors.
  * Patients with intolerance to salicylates.
  * Patients with verified, presumed or expected pregnancy or ongoing lactation.
  * Patients with liver cirrhosis, or evident hepatic or renal disease or insufficiency, and/or severe impairment of the bio-humoral parameters (i.e. 2 x upper limit of normal for alanine aminotransferase [ALT], aspartate aminotransferase [AST], gamma glutamyl transpeptidase [GGT] or creatinine).
  * Patient with severe diseases in other organs and systems.
  * Patients with local or systemic complications or other pathological states requiring a therapy with corticosteroids and/or immuno-suppressive agents.
  * Patients diagnosed with type 1 diabetes.
  * Patients diagnosed with, or with a family history of, glaucoma.
  * All patients with known hepatitis B, hepatitis C or with human immunodeficiency virus (HIV), according to the local privacy policy.
  * Participation in experimental therapeutic studies in the last 3 months. (Note: patients who participated in observational only studies are not excluded).
  * Any other medical condition that in the principal investigator's opinion would make the administration of the study drug or study procedures hazardous to the subject or obscure the interpretation of adverse events (AEs).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2008-06; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Eric Sands, Principal Investigator — Massachusetts General Hospital
Locations (105):
- United States (76):
  - Santarus Clinical Investigational Site 5051, Huntsville, Alabama
  - Santarus Clinical Investigational Site 5102, Mobile, Alabama
  - Santarus Clinical Investigational Site 5014, Sylacauga, Alabama
  - Santarus Clinical Investigational Site 5088, Tucson, Arizona
  - Santarus Clinical Investigational Site 5044, Anaheim, California
  - Santarus Clinical Investigational Site 5099, Encinitas, California
  - Santarus Clinical Investigational Site 5075, Fremont, California
  - Santarus Clinical Investigational Site 5087, Lakewood, California
  - Santarus Clinical Investigational Site 5033, Los Angeles, California
  - Santarus Clinical Investigational Site 5070, Palm Springs, California
  - Santarus Clinical Investigational Site 5067, San Diego, California
  - Santarus Clinical Investigational Site 5028, San Francisco, California
  - Santarus Clinical Investigational Site 5089, Boynton Beach, Florida
  - Santarus Clinical Investigational Site 5041, Hollywood, Florida
  - Santarus Clinical Investigational Site 5055, New Smyrna Beach, Florida
  - Santarus Clinical Investigational Site 5074, Port Orange, Florida
  - Santarus Clinical Investigational Site 5032, Tampa, Florida
  - Santarus Clinical Investigational Site 5009, Tampa, Florida
  - Santarus Clinical Investigational Site 5110, West Palm Beach, Florida
  - Santarus Clinical Investigational Site 5047, Winter Park, Florida
  - Santarus Clinical Investigational Site 5003, Zephyrhills, Florida
  - Santarus Clinical Investigational Site 5016, Atlanta, Georgia
  - Santarus Clinical Investigational Site 5056, Columbus, Georgia
  - Santarus Clinical Investigational Site 5103, Savannah, Georgia
  - Santarus Clinical Investigational Site 5085, Addison, Illinois
  - Santarus Clinical Investigational Site 5068, Evanston, Illinois
  - Santarus Clinical Investigational Site 5086, Bloomington, Indiana
  - Santarus Clinical Investigational Site 5053, Clive, Iowa
  - Santarus Clinical Investigational Site 5008, Metairie, Louisiana
  - Santarus Clinical Investigational Site 5090, Annapolis, Maryland
  - Santarus Clinical Investigational Site 5025, Baltimore, Maryland
  - Santarus Clinical Investigational Site 5092, Hollywood, Maryland
  - Santarus Clinical Investigational Site 5077, Prince Frederick, Maryland
  - Santarus Clinical Investigational Site 5046, Boston, Massachusetts
  - Santarus Clinical Investigational Site 5115, Brockton, Massachusetts
  - Santarus Clinical Investigational Site 5010, Chesterfield, Michigan
  - Santarus Clinical Investigational Site 5006, Troy, Michigan
  - Santarus Clinical Investigational Site 5004, Wyoming, Michigan
  - Santarus Clinical Investigational Site 5105, St Louis, Missouri
  - Santarus Clinical Investigational Site 5094, Egg Harbor, New Jersey
  - Santarus Clinical Investigational Site 5005, Marlton, New Jersey
  - Santarus Clinical Investigational Site 5024, Vineland, New Jersey
  - Santarus Clinical Investigational Site 5011, Great Neck, New York
  - Santarus Clinical Investigational Site 5101, New York, New York
  - Santarus Clinical Investigational Site 5020, Pittsford, New York
  - Santarus Clinical Investigational Site 5096, Fayetteville, North Carolina
  - Santarus Clinical Investigational Site 5058, Huntersville, North Carolina
  - Santarus Clinical Investigational Site 5091, New Bern, North Carolina
  - Santarus Clinical Investigational Site 5124, Wilmington, North Carolina
  - Santarus Clinical Investigational Site 5118, Canton, Ohio
  - Santarus Clinical Investigational Site 5045, Cincinnati, Ohio
  - Santarus Clinical Investigational Site 5078, Dayton, Ohio
  - Santarus Clinical Investigational Site 5120, Mentor, Ohio
  - Santarus Clinical Investigational Site 5066, Duncansville, Pennsylvania
  - Santarus Clinical Investigational Site 5065, Pottstown, Pennsylvania
  - Santarus Clinical Investigational Site 5035, Sayre, Pennsylvania
  - Santarus Clinical Investigational Site 5107, Sioux Falls, South Dakota
  - Santarus Clinical Investigational Site 5130, Jackson, Tennessee
  - Santarus Clinical Investigational Site 5095, Kingsport, Tennessee
  - Santarus Clinical Investigational Site 5021, Austin, Texas
  - Santarus Clinical Investigational Site 5076, Houston, Texas
  - Santarus Clinical Investigational Site 5108, Houston, Texas
  - Santarus Clinical Investigational Site 5019, Houston, Texas
  - Santarus Clinical Investigational Site 5036, Houston, Texas
  - Santarus Clinical Investigational Site 5063, Irving, Texas
  - Santarus Clinical Investigational Site 5072, Kingwood, Texas
  - Santarus Clinical Investigational Site 5054, La Porte, Texas
  - Santarus Clinical Investigational Site 5030, Lewisville, Texas
  - Santarus Clinical Investigational Site 5093, Plano, Texas
  - Santarus Clinical Investigational Site 5049, San Antonio, Texas
  - Santarus Clinical Investigational Site 5100, San Antonio, Texas
  - Santarus Clinical Investigational Site 5079, San Antonio, Texas
  - Santarus Clinical Investigational Site 5098, Tomball, Texas
  - Santarus Clinical Investigational Site 5015, Salt Lake City, Utah
  - Santarus Clinical Investigational Site 5097, Christiansburg, Virginia
  - Santarus Clinical Investigational Site 5119, Norfolk, Virginia
- Canada (10):
  - Santarus Clinical Investigational Site 6005, Abbotsford, British Columbia
  - Santarus Clinical Investigational Site 6000, Vancouver, British Columbia
  - Santarus Clinical Investigational Site 6014, Vancouver, British Columbia
  - Santarus Clinical Investigational Site 6008, Victoria, British Columbia
  - Santarus Clinical Investigational Site 6004, Richmond Hill, Ontario
  - Santarus Clinical Investigational Site 6017, Toronto, Ontario
  - Santarus Clinical Investigational Site 6001, Montreal, Quebec
  - Santarus Clinical Investigational Site 6002, Québec, Quebec
  - Santarus Clinical Investigational Site 6016, Saskatoon, Saskatchewan
  - Santarus Clinical Investigational Site 6006, Toronto
- India (18):
  - Santarus Clinical Investigational Site 9001, Andhra Pradesh
  - Santarus Clinical Investigational Site 9009, Andhra Pradesh
  - Santarus Clinical Investigational Site 9012, Andhra Pradesh
  - Santarus Clinical Investigational Site 9016, Andhra Pradesh
  - Santarus Clinical Investigational Site 9006, Assam
  - Santarus Clinical Investigational Site 9007, Gujarat
  - Santarus Clinical Investigational Site 9004, Karnataka
  - Santarus Clinical Investigational Site 9015, Karnataka
  - Santarus Clinical Investigational Site 9003, Kerala
  - Santarus Clinical Investigational Site 9002, Maharashtra
  - Santarus Clinical Investigational Site 9008, Maharashtra
  - Santarus Clinical Investigational Site 9010, Maharashtra
  - Santarus Clinical Investigational Site 9011, Maharashtra
  - Santarus Clinical Investigational Site 9013, Maharashtra
  - Santarus Clinical Investigational Site 9017, Maharashtra
  - Santarus Clinical Investigational Site 9018, Rajasthan
  - Santarus Clinical Investigational Site 9005, Tamil Nadu
  - Santarus Clinical Investigational Site 9014, Uttar Pradesh
- Santarus Clinical Investigational Site 7000, Central, La Paz Baja California Sur, Mexico

REFERENCES:
- [Result] Sandborn WJ, Travis S, Moro L, Jones R, Gautille T, Bagin R, Huang M, Yeung P, Ballard ED 2nd. Once-daily budesonide MMX(R) extended-release tablets induce remission in patients with mild to moderate ulcerative colitis: results from the CORE I study. Gastroenterology. 2012 Nov;143(5):1218-1226.e2. doi: 10.1053/j.gastro.2012.08.003. Epub 2012 Aug 11. PMID 22892337

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from August 2008 until May 2010.
Pre-assignment Details: Diary data for symptoms will be collected prior to randomization. Lab testing and a colonoscopy will be done prior to randomization. 510 patients were randomized. One patient was not treated and was not included in baseline characteristics, efficacy, and safety analyses. 509 patients received study drug and were included in safety analyses.
Groups:
- 1: Budesonide-MMX® 6 mg: One budesonide-MMX® 6 mg plus two placebo Asacol® overencapsulated tablets daily in the morning after breakfast and two placebo Asacol® overencapsulated tablets daily after the mid-day meal and the evening meal for eight weeks.
  budesonide-MMX® 6 mg : 6 mg/day, 6 mg tablets
  Blood sampling, endoscopy : Blood sampling for hematology and biochemistry and endoscopy with biopsy for histological and endoscopic assessment scores
- 2: Budesonide-MMX® 9 mg: One budesonide-MMX® 9 mg plus two placebo Asacol® overencapsulated tablets daily in the morning after breakfast and two placebo Asacol® overencapsulated tablets daily after the mid-day meal and the evening meal for eight weeks.
  Blood sampling, endoscopy : Blood sampling for hematology and biochemistry and endoscopy with biopsy for histological and endoscopic assessment scores
  budesonide-MMX® 9 mg : 9 mg/day, 9 mg tablets
- 3: Placebo: Two placebo Asacol® overencapsulated tablets plus one placebo Budesonide MMX® tablet daily in the morning after breakfast and two placebo Asacol® overencapsulated tablets daily after the mid-day meal and the evening meal for eight weeks.
  Placebo : Placebo
  Blood sampling, endoscopy : Blood sampling for hematology and biochemistry and endoscopy with biopsy for histological and endoscopic assessment scores
- 4: Asacol® 400 mg: Two Asacol® 400 mg overencapsulated tablets plus one placebo budesonide MMX® tablet daily in the morning after breakfast and two Asacol® 400 mg overencapsulated tablets daily after the mid-day meal and the evening meal for eight weeks.
  Asacol® 400 mg : 2400 mg/day, 400 mg tablets
  Blood sampling, endoscopy : Blood sampling for hematology and biochemistry and endoscopy with biopsy for histological and endoscopic assessment scores
Period: Overall Study
Arm/Group | 1: Budesonide-MMX® 6 mg | 2: Budesonide-MMX® 9 mg | 3: Placebo | 4: Asacol® 400 mg
Started | 126 | 127 | 129 | 127
Completed | 89 | 89 | 76 | 95
Not Completed | 37 | 38 | 53 | 32
Not completed — Adverse Event | 5 | 6 | 10 | 7
Not completed — Protocol Violation | 1 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 8 | 11 | 10 | 9
Not completed — Lost to Follow-up | 1 | 5 | 4 | 2
Not completed — Physician Decision | 3 | 2 | 2 | 2
Not completed — Sponsor decision | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 13 | 9 | 14 | 8
Not completed — Infectious colitis, normal histology | 5 | 4 | 8 | 3
Not completed — Randomization error, return to prior Rx | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population= primary population for efficacy/baseline characteristics analyses. ITT population= randomized patients who received study drug, and did not include patients with major entry criteria/GCP violations or normal histology at baseline (N= 509 randomized - 3[infectious colitis] - 17[normal histology at baseline] = 489).
Groups:
- Total: Total of all reporting groups
Arm/Group | 1: Budesonide-MMX® 6 mg | 2: Budesonide-MMX® 9 mg | 3: Placebo | 4: Asacol® 400 mg | Total
Number analyzed (Participants) | 121 | 123 | 121 | 124 | 489
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 117 | 122 | 115 | 118 | 472
  >=65 years | 4 | 1 | 6 | 6 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (13) | 41.7 (12.2) | 41.7 (13.6) | 44 (12.4) | 42.7 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 46 | 53 | 55 | 216
  Male | 59 | 77 | 68 | 69 | 273
Region of Enrollment [Number; unit: participants]
  United States | 75 | 76 | 77 | 76 | 304
  Canada | 5 | 7 | 5 | 6 | 23
  India | 41 | 40 | 39 | 42 | 162

OUTCOME MEASURES:

1. Primary Outcome: Clinical and Endoscopic Remission.
Description: Clinical and endoscopic remission defined as a Ulcerative Colitis Disease Activity Index (UCDAI) score ≤ 1, with subscores of 0 for rectal bleeding, stool frequency, and mucosal appearance and with a ≥ 1 point reduction in the endoscopic index score.
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | 1: Budesonide-MMX® 6 mg | 2: Budesonide-MMX® 9 mg | 3: Placebo | 4: Asacol® 400 mg
Number analyzed (Participants) | 121 | 123 | 121 | 124
percentage of patients | 13.2 [7.2 to 19.3] | 17.9 [11.1 to 24.7] | 7.4 [2.8 to 12.1] | 12.1 [6.4 to 17.8]
Statistical Analysis 1: Comparison: 1: Budesonide-MMX® 6 mg vs 3: Placebo; All p-values were based on the Chi-square test; comparisons of budesonide MMX and placebo were conducted at the α = 0.025 level of significance and the comparison of Asacol and placebo were conducted at the α = 0.05 level of significance. The study was not powered to show statistical significance for Asacol versus budesonide MMX; Test type: Superiority or Other; p = 0.1393, Chi-squared; Difference in proportions = 5.8, 95% CI 2-sided [-1.8 to 13.4] — The difference in proportions was determined by subtracting the proportion of patients who reached the endpoint in the placebo group from that proportion in the active group (active minus placebo)
Statistical Analysis 2: Comparison: 2: Budesonide-MMX® 9 mg vs 3: Placebo; See comments from the budesonide 6 mg versus placebo comparison (statistical analysis 1); Test type: Superiority or Other; p = 0.0143, Chi-squared; Difference in proportions = 10.4, 95% CI 2-sided [2.2 to 18.7] — See comments from the budesonide 6 mg versus placebo comparison (statistical analysis 1)
Statistical Analysis 3: Comparison: 3: Placebo vs 4: Asacol® 400 mg; See comments from the budesonide 6 mg versus placebo comparison (statistical analysis 1); Test type: Superiority or Other; p = 0.2200, Chi-squared; Difference in proportions = 4.7, 95% CI 2-sided [-2.7 to 12.1] — See comments from the budesonide 6 mg versus placebo comparison (statistical analysis 1)

2. Secondary Outcome: Clinical Improvement.
Description: Clinical improvement, defined as a ≥ 3-point improvement in UCDAI from baseline to the end of Week 8.
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | 1: Budesonide-MMX® 6 mg | 2: Budesonide-MMX® 9 mg | 3: Placebo | 4: Asacol® 400 mg
Number analyzed (Participants) | 121 | 123 | 121 | 124
percentage of patients | 30.6 [22.4 to 38.8] | 33.3 [25.0 to 41.7] | 24.8 [17.1 to 32.5] | 33.9 [25.5 to 42.2]
Statistical Analysis 1: Comparison: 1: Budesonide-MMX® 6 mg vs 3: Placebo; Clinical improvement and endoscopic improvement were analyzed hierarchically. If at least one primary endpoint comparison was statistically significant, clinical improvement was to be compared between each budesonide MMX group and placebo at the α = 0.025 level of significance. If at least one comparison of clinical improvement was statistically significant, endoscopic improvement was to be compared between each budesonide MMX dose group and placebo at the α = 0.025 level of significance; Test type: Superiority or Other; p = 0.3146, Chi-squared; Difference in proportions = 5.8, 95% CI 2-sided [-5.5 to 17.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 2: Budesonide-MMX® 9 mg vs 3: Placebo; See comments from the budesonide 6 mg versus placebo comparison (statistical analysis 1); Test type: Superiority or Other; p = 0.1420, Chi-squared; Difference in proportions = 8.5, 95% CI 2-sided [-2.8 to 19.9] — See comments from the budesonide 6 mg versus placebo comparison (statistical analysis 1)
Statistical Analysis 3: Comparison: 3: Placebo vs 4: Asacol® 400 mg; See comments from the budesonide 6 mg versus placebo comparison (statistical analysis 1); Test type: Superiority or Other; p = 0.1189, Chi-squared; Difference in proportions = 9.1, 95% CI 2-sided [-2.3 to 20.4] — See comments from the budesonide 6 mg versus placebo comparison (statistical analysis 1)

3. Secondary Outcome: Endoscopic Improvement
Description: Greater or equal to a 1 point improvement in the mucosal appearance subscore of the UCDAI, from baseline to week 8.
  As per the hierarchical testing procedure for secondary endpoints, because clinical improvement was not statistically significant in the ITT population, formal statistical comparisons for endoscopic improvement between the 2 budesonide MMX groups and placebo were not conducted.
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | 1: Budesonide-MMX® 6 mg | 2: Budesonide-MMX® 9 mg | 3: Placebo | 4: Asacol® 400 mg
Number analyzed (Participants) | 121 | 123 | 121 | 124
percentage of patients | 35.5 [27 to 44.1] | 41.5 [32.8 to 50.2] | 33.1 [24.7 to 41.4] | 33.1 [24.8 to 41.3]
Statistical Analysis 1: Comparison: 3: Placebo vs 4: Asacol® 400 mg; As per the hierarchical testing procedure for secondary endpoints, because clinical improvement was not statistically significant in the ITT population, formal statistical comparisons for endoscopic improvement between the 2 budesonide MMX groups and placebo were not conducted. The statistical comparison between the Asacol and placebo groups is shown here; Test type: Superiority or Other; p = 0.9991, Chi-squared; Difference in proportions = 0.0, 95% CI 2-sided [-11.8 to 11.8] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 56 day ± 2 day (study duration) + 30 day safety followup period.
Description: Adverse event data were analyzed using the safety population, defined as all patients who received study drug. 509 patients received study drug and were included in safety analyses.
Arm/Group | 1: Budesonide-MMX® 6 mg | 2: Budesonide-MMX® 9 mg | 3: Placebo | 4: Asacol® 400 mg
Serious Adverse Events (participants affected / at risk) | 2/126 | 3/127 | 3/129 | 4/127
Other Adverse Events (participants affected / at risk) | 35/126 | 36/127 | 34/129 | 31/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1: Budesonide-MMX® 6 mg (N=126) | 2: Budesonide-MMX® 9 mg (N=127) | 3: Placebo (N=129) | 4: Asacol® 400 mg (N=127)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1: Budesonide-MMX® 6 mg (N=126) | 2: Budesonide-MMX® 9 mg (N=127) | 3: Placebo (N=129) | 4: Asacol® 400 mg (N=127)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 4 (4) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 2 (3) | 4 (6) | 2 (2) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 6 (7) | 8 (9) | 10 (10)
Abdominal pain upper (Gastrointestinal disorders) | 5 (8) | 5 (7) | 2 (3) | 2 (3)
Abdominal tenderness (Gastrointestinal disorders) | 3 (5) | 1 (1) | 2 (2) | 3 (3)
Colitis ulcerative (Gastrointestinal disorders) | 15 (15) | 12 (12) | 20 (20) | 12 (12)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 1 (1) | 7 (7) | 8 (9)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (2) | 4 (4) | 5 (6)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (3) | 7 (7)
Frequent bowel movements (Gastrointestinal disorders) | 2 (3) | 1 (1) | 3 (4) | 4 (5)
Nausea (Gastrointestinal disorders) | 5 (6) | 5 (5) | 8 (10) | 10 (10)
Vomiting (Gastrointestinal disorders) | 5 (5) | 0 (0) | 4 (4) | 3 (5)
Asthenia (General disorders) | 4 (5) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 3 (3) | 5 (5) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 5 (6) | 3 (4) | 9 (9) | 3 (3)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (5) | 3 (3) | 4 (4) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 2 (2) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 5 (5) | 1 (1) | 3 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Blood cortisol decreased (Investigations) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 2 (2) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5) | 7 (9) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 4 (8) | 2 (3)
Dizziness (Nervous system disorders) | 6 (7) | 0 (0) | 1 (1) | 4 (5)
Headache (Nervous system disorders) | 17 (29) | 8 (14) | 19 (31) | 12 (15)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 6 (8) | 5 (5) | 9 (10) | 3 (4)
Mood altered (Psychiatric disorders) | 4 (5) | 2 (2) | 2 (2) | 3 (3)
Pollakiuria (Renal and urinary disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (5) | 2 (2) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 5 (6) | 3 (4)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No